CLINICAL TRIAL: NCT00247975
Title: Primary Prevention of Anthracycline-Induced Cardiotoxicity With L-Carnitine in Patients With Breast Cancer (PPACC)-Pilot Study
Brief Title: Ability of L-carnitine to Prevent Heart Damage in Breast Cancer Patients Receiving Anthracycline Chemotherapy
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Insufficient recruitment
Sponsor: Ottawa Heart Institute Research Corporation (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: CIHR #: 126541
Record Dates: First submitted 2005-10-31; First posted 2005-11-02 (Estimated); Last update posted 2022-08-16 (Actual); Status verified 2022-08

CONDITIONS: Heart Failure
Keywords: L-carnitine; Breast cancer; Anthracycline Cardiotoxicity; Primary prevention; Anthracycline induced cardiotoxicity; Left Ventricular Ejection Fraction
MeSH Terms: conditions — Heart Failure; Breast Neoplasms | interventions — Carnitine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: L-carnitine — Patients will be randomized to L-carnitine therapy or placebo. Patients in the treatment group will receive oral L-carnitine (3 grams daily) for 3 days prior to chemotherapy, 1 gram of intravenous L-carnitine (5 cc over 5 minutes, prior to chemotherapy) on the day of chemotherapy and oral L-carnitine (3 grams daily) for 3 days after chemotherapy.
  Other Names: Sigma-Tau

SUMMARY:
Breast cancer is very common and afflicts 1 in 9 North American women. The treatment of breast cancer often requires the use of chemotherapy including "anthracyclines". Anthracyclines can damage the heart resulting in heart failure and even death. Clinicians and researchers are continually seeking methods that will reduce the toxic effects of anthracycline treatment.

L-carnitine is a substance that is produced naturally in the body and is required for normal heart function. Animal studies have suggested that L-carnitine protects the heart from the effects of anthracyclines, however this has not been verified in humans.

This study will assess the potential role of L-carnitine in the prevention of anthracycline induced heart damage. The investigators will enroll 144 patients into this study. Patients will be randomly assigned to L-carnitine therapy or to standard care (no L-carnitine therapy). Patients in the L-carnitine group will receive oral and intravenous L-carnitine prior to and after their anthracycline therapy. Patients will undergo regular follow up and testing to assess heart function. The investigators believe that patients treated with L-carnitine will benefit and have fewer complications associated with anthracycline treatment.

ELIGIBILITY:
Inclusion Criteria:

* Female patients must have histologically or cytologically indicated breast cancer (stages I, II, III) eligible for adjuvant anthracycline chemotherapy [FEC100 or AC-Taxol(paclitaxel) every 21 days.
* HER2 negative or HER2 positive breast cancer by immunohistochemistry (IHC3+) and/or fluorescent in-situ hybridization.
* Eastern cooperative oncology group (ECOG) performance status = 0, 1, 2
* Age ≥ 18 years old.
* Ability to understand and the willingness to sign a written informed consent document.
* The effects of L-carnitine on the developing human fetus at the recommended therapeutic dose are unknown. For this reason, women of child-bearing potential must agree to use adequate contraception prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately.

Exclusion Criteria:

* Patients with evidence of metastatic breast cancer.
* Resting LV ejection fraction < 50%.
* Patients having received previous anthracycline therapy or contraindication to anthracycline.
* Patients having a contraindication to L-carnitine therapy
* Dexrazoxane therapy at the time of enrollment.
* Patients with abnormal baseline bloodwork:

  * hemoglobin ≤ 100 mg/L
  * platelets ≤ 100 x 10^9/L
  * white blood cells ≤ 4 x 10^9/L
  * creatinine, AST, ALT, bilirubin > 1.5 x the upper normal limits
* Participation in another randomized clinical trial.
* Patients having significant cardiac disease (previous myocardial infarction, congestive heart failure, or hemodynamically significant valvular heart disease) that would limit compliance with study requirements.
* Patients taking medication that may affect LV function (b-blockers, amiodarone, ACE-inhibitors, calcium channel blockers, or digoxin).
* Patients with symptoms of heart failure.
* Patients unable to participate in a study requiring long term follow up.
* Pregnant or lactating women.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2006-03; Primary Completion 2010-10 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
To compare the effects of L-carnitine therapy versus placebo on left ventricular (LV) ejection fraction (EF) as a marker of anthracycline induced cardiotoxicity | 1 year

SECONDARY OUTCOMES:
To compare the effects of L-carnitine therapy versus placebo on: other potential markers of anthracycline induced cardiotoxicity such as LV volume, LV systolic and diastolic function, troponin T (TnT) and NT-pro-brain natriuretic peptide (BNP) | 1 year
"Anthracycline-induced cardiotoxicity" and clinical cardiac outcomes | 1 year
Serum L-carnitine levels | 4 months
To assess: the safety of L-carnitine | 1 year
the predictive value of serum biomarkers (TnT, BNP, and L-carnitine levels) for cardiotoxicity and cardiac outcome (ejection fraction, LV volumes, congestive heart failure, and cardiac death) | 1 year
the effect of anthracyclines on plasma L-carnitine levels | 4 months
the correlation of L-carnitine levels with serum TnT and BNP levels | 4 months

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin JW Chow, MD, FRCPC, Principal Investigator — Ottawa Heart Institute Research Corporation; Rob S Beanlands, MD, FRCPC, Study Chair — Ottawa Heart Institute Research Corporation; Haissam Haddad, MD, FRCPC, Study Chair — Ottawa Heart Institute Research Corporation; George Wells, M.Sc., PhD, Study Chair — Ottawa Heart Institute Research Corporation; Susan Dent, MD, FRCPC, Study Chair — Ottawa Regional Cancer Centre; Sean Hopkins, B.Sc, RPEBC, Study Chair — Ottawa Regional Cancer Centre; Michele A Turek, MD, FRCPC, Study Chair — Ottawa Hospital
Locations (1):
- University of Ottawa Heart Institute, Ottawa, Ontario, Canada